CLINICAL TRIAL: NCT03091985
Title: Influence of the Brownie Breast Shield on the Dynamics of Milk Removal
Acronym: BDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medela AG (Industry)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: MHM1601
Record Dates: First submitted 2017-03-15; First posted 2017-03-27 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2018-02

CONDITIONS: Lactation
Keywords: Breastshield; Breastpump; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Drainage of the lactating breast using:
  PersonalFit - Breast shield & Brownie - Breast shield
  Breast shields are each to be used for 15 min pumping with the symphony breastpump
  Interventions: Device: PersonalFit - Breast shield; Device: Brownie - Breast shield
- Group B (Experimental): Drainage of the lactating breast using:
  Brownie - Breast shield & PersonalFit - Breast shield
  Breast shields are each to be used for 15 min pumping with the symphony breastpump
  Interventions: Device: PersonalFit - Breast shield; Device: Brownie - Breast shield

INTERVENTIONS:
Device: PersonalFit - Breast shield — Subjects are to pump 15 min with the comparator device
Device: Brownie - Breast shield — Subjects are to pump 15 min with the investigational device

SUMMARY:
The purpose of this study is to investigate the efficacy of breast drainage of the healthy breast with the new Medela pump set breast shield (Brownie).

The objective of the study is to verify the Brownie breast shield to be non-inferior to the current PersonalFit breast shield in emptying the healthy lactating breast.

DETAILED DESCRIPTION:
In this study we could show that the Brownie shield is non-inferior to the PersonalFit shield in all four endpoints, superior to the PersonalFit shield in terms of PAMR and expressed milk volume, and is more comfortable than the PersonalFit shield according to participant surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years old
2. Infant is ≥1 and ≤6 month old
3. Subject is predominantly breastfeeding (80% of all feeds, i.e. ≤150 ml formula/day or equal representative amount of solid food)
4. The subject agrees to pump or feed the last time a minimum of 3 hours before the start of the pumping session at the study site
5. The subject agrees to photographs of the breast and upper body (no face)
6. The subject agrees to perform a 24 hour milk production at home, inclusive weighing the Infant before and after each feeding
7. The subject agrees to collect ~2 ml of milk before and after each feeding for fat analysis
8. The subject signed the Informed Consent Form

Exclusion Criteria:

1. Mastitis (any breast within two weeks prior enrolment)
2. Engorgement (any breast within two weeks prior enrolment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the nature of the study device (breastshiled to be used for expressing breastmilk) only lactating females can be enrolled into the study.
Enrollment: 49 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
PAMR | 7-21 days
  Breast drainage, determined by the metric percent of available milk removed (PAMR).

SECONDARY OUTCOMES:
Milk volume | After 15 minutes of controlled pumping with the test or comparator device. Each participant will pump twice with a "washout period" of 7-21 days in between the corresponding occasions.
  Expressed breast milk volume
Mid fat content | After 15 minutes of controlled pumping with the test or comparator device. Each participant will pump twice with a "washout period" of 7-21 days in between the corresponding occasions.
  Breast milk - mid fat content
Hind fat content | After 15 minutes of controlled pumping with the test or comparator device. Each participant will pump twice with a "washout period" of 7-21 days in between the corresponding occasions.
  Breast milk - hind fat content
Device usability | After 15 minutes of controlled pumping with the test or comparator device. Each participant will pump twice with a "washout period" of 7-21 days in between the corresponding occasions.
  Device usability questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Ivarsson, PhD, Principal Investigator — Employee
Locations (1):
- Medela AG, Baar, Canton of Zug, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sakalidis VS, Ivarsson L, Haynes AG, Jager L, Scharer-Hernandez NG, Mitoulas LR, Prime DK. Breast shield design impacts milk removal dynamics during pumping: A randomized controlled non-inferiority trial. Acta Obstet Gynecol Scand. 2020 Nov;99(11):1561-1567. doi: 10.1111/aogs.13897. Epub 2020 Jun 5. PMID 32401335